CLINICAL TRIAL: NCT03590002
Title: A Cluster-specific Pre-post Trial With Randomized and Staggered Implementation to Evaluate the Effectiveness of an Electronic ICU Medical Transfer of Care Document to Improve Communication During ICU-to-Ward Transfers of Care
Brief Title: Evaluating the Effectiveness of an Electronic Medical Transfer Tool to Improve Communication During Transfers From ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry T. Stelfox, MD PhD (Other)
Collaborators: Canadian Frailty Network (Other); Alberta Health services (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Henry T. Stelfox, MD PhD, Professor, University of Calgary
Organization: University of Calgary (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-2317
Record Dates: First submitted 2018-05-29; First posted 2018-07-18 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Critical Illness; Transitions of Care
Keywords: Patient Transfer; Patient Discharge Summaries; Continuity of Patient Care; Intensive Care Unit; Critical Care; Health Information Exchange; Medical Order Entry Systems; Point-of-Care Systems; Medical Informatics
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: All study ICUs will begin as control sites (i.e., no electronic medical transfer tool available). ICUs will be randomly allocated to cross over to the intervention (i.e., electronic medical transfer tool available) at regular intervals (approximately every eight weeks) until all ICUs receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic ICU Medical Transfer Tool (Experimental): ICUs allocated to the experimental arm will have access to the electronic Medical Transfer of Care Documentation Tool within the clinical information system (CIS) in order to prepare ICU transfer of care documents for the receiving medical care team.
  Interventions: Device: Electronic ICU Medical Transfer Tool
- Dictated ICU Medical Transfer (No Intervention): Usual Care, ICUs in the control group will only have access to the dictation documentation system as the standard method to prepare ICU medical transfer documents. New ICU medical staff responsible for preparing transfer documents will receive the usual training on the dictation system.

INTERVENTIONS:
Device: Electronic ICU Medical Transfer Tool — Patient transfers of care from the ICU to inpatient wards prepared using the electronic ICU medical transfer tool within the health zone's clinical information system, Sunrise Clinical Manager.
  Other Names: ICU Transfer Tool; ICU Medical Transfer Summary
  Arms: Electronic ICU Medical Transfer Tool

SUMMARY:
The transfer of patients from the intensive care unit (ICU) to a medical or surgical hospital ward is a particularly high risk transfer that may expose patients to complications or adverse events if there are communication breakdowns between sending and receiving medical teams. Current dictation practice often falls short in producing optimal clinical documentation on patients being transferred from the ICU to the ward. The use of an electronic transfer of care tool to standardize communication may improve the quality of information exchanged between ICU and ward medical teams during ICU transfers, compared to dictation. This study will stagger implementation of a new electronic ICU medical transfer of care tool across four adult medical-surgical ICUs in one city. It is anticipated that the electronic ICU transfer tool will positively impact two inter-related goals: (1) improve the completeness and timeliness of clinical documentation on transfer, and (2) reduce the incidence of associated adverse patient clinical outcomes after transfer (e.g., adverse events, ICU readmission).

DETAILED DESCRIPTION:
Background: Transfers of care within hospital are vulnerable periods in health care delivery. The complete, accurate, and timely communication of essential patient information is particularly critical in transfers of care from the intensive care unit (ICU) to an inpatient ward. The ICU generally has the most vulnerable patients, the highest resource use, and most complex system of multi professional coordinated care within the hospital. Communication breakdowns between ICU and receiving inpatient medical teams can have profound implications on the quality, delivery and cost of patient care. Ineffective transfers may result in adverse events, redundant testing, increased hospital stays, and readmission to ICU or hospital.

The written transfer summary is a widely used and important means to present and prioritize patient information to healthcare providers. Unlike verbal reporting, written communication is durable and accessible to many providers at many points in time, making it a critical component in facilitating continuity of patient care. Despite known shortcomings, dictation remains standard practice in many hospitals to complete ICU medical transfer summaries. Although the optimal content and structure for transfer summaries have not been agreed upon in the scientific community, it is clear that standardization can help minimize both the incidence and impact of information gaps during transfer. Computer-enabled tools that remind and guide the user to document essential content (e.g., goals of care, medications) have been found to improve the relevance, consistency, and readability of information in transfer summaries.

Methods: This study will use a cluster-specific pre-post trial design with randomized and staggered implementation to assess the effectiveness of an electronic transfer of care tool developed in the primary clinical information system (Sunrise Clinical Manager, Eclipsys Corporation, Boca Raton, FL) by a multidisciplinary team of healthcare providers and clinical documentation specialists. Four adult medical surgical ICUs in one Canadian city will begin as control sites (i.e., no electronic medical transfer tool available) and subsequently be allocated in a random order to cross over to intervention sites (i.e., electronic medical transfer tool available) at regular intervals. Implementation intervals will be matched to medical resident rotation block dates, which occur every four weeks; a single study interval will encompass two resident blocks. Users--physicians and nurse practitioners responsible for completing ICU medical transfer summaries--will have access to the electronic medical transfer tool at intervention sites, in addition to standard dictation services. A multi-component knowledge translation (KT) strategy designed to facilitate adoption of the tool will be tailored and delivered to ICUs prior to implementation at the site. The KT strategy will encompass education, point-of-care support, and audit and feedback.

Data will be collected both prospectively and retrospectively to measure perceived (prospective user survey) and actual (retrospective chart review) quality of the transfer summaries. The primary outcome will be a binary composite measure of two transfer summary conditions, manually collected retrospectively: (1) presence of four essential information elements (goals of care designation, diagnosis, active issues on transfer, medications to continue) and (2) availability of the transfer summary to accepting clinicians at the time of patient transfer. Transfer summaries that meet these two conditions will be coded as "Present"; those that do not will be coded as "Absent". Patient clinical outcome data also will be retrospectively collected from hospital clinical information systems and paper charts. All study outcomes will be compared between baseline (pre-implementation) and intervention (post-implementation) periods for all ICUs.

Discussion: The evaluation of the electronic medical ICU transfer tool will contribute to our understanding how computer-based structured documentation can improve communication between medical teams and potentially better patient safety.

ELIGIBILITY:
Inclusion Criteria:

* medical-surgical ICU patient
* ICU disposition on transfer is 'alive'
* Transfer to another patient care unit

Exclusion Criteria:

* ICU discharge to home/community residence
* ICU discharge by death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1751 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Complete and Timely ICU medical transfer of care document | Day 1, post patient ICU discharge
  Binary measure of the presence/absence of two conditions (1) presence of four essential information elements in ICU transfer document (GOC designation, diagnosis, active health issues, and active medications), and (2) availability of the document to accepting medical team at the time of patient transfer. Both conditions must be met to be coded as present.

SECONDARY OUTCOMES:
Overall completeness of ICU medical transfer of care document | Day 1, post patient ICU-discharge
  Composite measure of presence of eight essential information fields in ICU transfer document
Timeliness of ICU medical transfer of care document | Day 1, post patient ICU discharge
  Availability of ICU transfer of care document in the clinical information system
Quality Ratings of ICU clinicians | 2 year
  ICU clincian ratings of a sample of transfer of care documents.
Adverse Event | Post patient ICU discharge, up to 72 hours
  Adverse Event is defined as an injury or harm related to (or from) the delivery of care. A two-stage manual abstraction process based on the Institute for Healthcare Improvement Global Trigger Tool (GTT) method of chart review will be applied retrospectively to a random sample of patients.
Perceptions of ICU clinicians | 2 year
  Survey of ICU clinicians on preparing transfer of care document and perceptions of quality.

OTHER OUTCOMES:
ICU Readmission | Post patient ICU discharge, up to 72 hours
  Patient readmission to ICU after having been previously transferred from ICU to ward
Medical Emergency Team (MET) Activation | Post patient ICU discharge, up to 72 hours
  Patient experienced sudden clinical deterioration that triggered MET activation
Cardiac Arrest Event | Post patient ICU discharge, up to 72 hours
  Patient experienced a cardiac arrest event as recorded in hospital system by Code Blue team
Hospital Mortality | Post patient ICU discharge, up to 60 days
  Patient died within hospital after ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Henry T Stelfox, MD, PhD, Principal Investigator — University of Calgary; Jeanna Parsons Leigh, PhD, Principal Investigator — Dalhouse University
Locations (4):
- Canada (4):
  - Intensive Care Unit, Peter Lougheed Centre, Calgary, Alberta
  - Intensive Care Unit, Foothills Medical Centre, Calgary, Alberta
  - Intensive Care Unit, Rockyview General Hospital, Calgary, Alberta
  - Intensive Care Unit, South Health Campus, Calgary, Alberta

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data will be uploaded into the primary funding agency, Canadian Frailty Network (CFN), digital data management system (DDMS) which is currently being developed by the CFN.
Supporting Information: Study Protocol, SAP
Time Frame: To be determined once the DDMS is developed.
Access Criteria: To be determined once the DDMS is developed.

REFERENCES:
- [Background] Parsons Leigh J, Brundin-Mather R, Zjadewicz K, Soo A, Stelfox HT. Improving transitions in care from intensive care units: Development and pilot testing of an electronic communication tool for healthcare providers. J Crit Care. 2020 Apr;56:265-272. doi: 10.1016/j.jcrc.2020.01.019. Epub 2020 Jan 18. No abstract available. PMID 31986370
- [Background] Parsons Leigh J, Brundin-Mather R, Whalen-Browne L, Kashyap D, Sauro K, Soo A, Petersen J, Taljaard M, Stelfox HT. Effectiveness of an Electronic Communication Tool on Transitions in Care From the Intensive Care Unit: Protocol for a Cluster-Specific Pre-Post Trial. JMIR Res Protoc. 2021 Jan 8;10(1):e18675. doi: 10.2196/18675. PMID 33416509